CLINICAL TRIAL: NCT04977362
Title: Interdisciplinary and Cross-sectoral Perioperative Care Model in the Cardiac Surgery: Implementation in the Setting of Minimally-invasive Heart Valve Surgery (INCREASE)
Brief Title: Interdisciplinary Perioperative Care in Minimally-invasive Heart Valve Surgery
Acronym: INCREASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: BARMER (Other); University Hospital Augsburg (Other)
Responsible Party: Principal Investigator, Evaldas Girdauskas, Prof. Dr. med., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1564/108
Record Dates: First submitted 2021-06-18; First posted 2021-07-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Heart Valve Diseases
Keywords: randomized controlled trial; enhanced recovery after surgery; minimally invasive surgery; postanesthesia care unit; physiotherapy
MeSH Terms: conditions — Heart Valve Diseases | interventions — Enhanced Recovery After Surgery; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator
Masking Description: All scientists and statisticans involved in the analysis of the study will be blinded to the allocation of participants and will receive only pseudomized data from the study coordinator, who organises data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS protocol (intervention group) (Experimental): The innovative care process in the intervention group is characterized by an interdisciplinary approach according to the previously established enhanced recovery after surgery protocol. This process aims at improving the clinical outcome after cardiac surgery, increasing patient satisfaction and quality of life, enabling early professional reentry and participation, and optimizing the cost-effectiveness of service provision. In addition, intersectoral barriers are being broken down in order to establish an interdisciplinary and cross-sectoral overall care process for patients with heart valve surgery as a new form of care in the future.
  Interventions: Other: Enhanced Recovery After Surgery
- Treatment as usual (control group) (Active Comparator): The control group undergoes standard heart valve surgery. In this case, no preoperative interventions take place, the patient is operated on the affected heart valve in a minimally invasive procedure without prehabilitation. After surgery, the patient is transfered to an intensive care unit (not a specialized postanesthesia care unit) depending on the individual condition and then transfered to the general ward. Patients receive medical, nursing, and physiotherapeutic care in accordance with current hospital standards.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Enhanced Recovery After Surgery — Enhanced recovery after surgery is a multimodal, transdisciplinary care approach for patients undergoing surgical procedures. It is implemented in various surgical specialties, among others in cardiac surgery. The care approach aims at promotion of recovery of the patients throughout their perioperative process, reduction of complications, and early return to normal activities.
  Other Names: fast track; rapid recovery; ERAS
  Arms: ERAS protocol (intervention group)
Other: Treatment as Usual — treatment as usual according to standard care in heart valve surgery
  Arms: Treatment as usual (control group)

SUMMARY:
Valvular heart diseases are among the most common cardiac pathologies in adult patients in Germany. Currently, the process of care before, during and after heart valve surgery does not follow a standardized and interdisciplinary optimal approach. An approach already established in other surgical disciplines is the Enhanced Recovery After Surgery (ERAS) protocol, which aims at optimizing the recovery process of patients. Within the INCREASE study, a care process inspired by the ERAS protocol will be established at the University Heart and Vascular Center (UHZ) of the University Medical Center Hamburg-Eppendorf (UKE) and the University Medical Center Augsburg (UKA). Executing the study at two facilities in different regions in Germany will help to demonstrate transferability of the process of care. The effectiveness of this process compared to the current treatment approach will be investigated in a randomized controlled trial. A total of 186 patients will be allocated by chance either to the intervention group (ERAS protocol) or the control group (treatment as usual). Patients in the intervention group will receive an optimized interdisciplinary care protocol including medical, nursing, physiotherapeutical and psychotherapeutical interventions. Measurements of effectiveness are the number of hospitalized days (due to cardiac causes) within one year and the physical condition of the patient as measured by the 6-minute walk test (6MWT) on the day of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective minimally invasive (open) aortic or mitral valve surgery
* Patient's ability to understand the nature and extent of the individual's requirements for participation in the new care setting
* Classification of the patient as "FIT" or "Pre-FRAIL" using the LUCAS functional index (frailty index) (Dapp et al. 2012)

Exclusion Criteria:

* Limited life expectancy less than one year (e.g., advanced tumor disease)
* Urgent or emergency interventions
* Severe chronic obstructive pulmonary disease (GOLD III or IV)
* Dialysis-dependant renal failure
* Advanced liver cirrhosis (Child stages B + C)
* Severe comorbidities or psychosocial reasons that militate against participation or do not allow for written informed consent (e. g., residual neurological impairment after prior stroke, major restrictions of mobility, neuropsychological disorders, depressive disorder, substance-related addictive disorders)
* Lack of a social environment that can provide supportive patient care
* Previous cardiac surgery (i.e., relative contraindication for minimally invasive technique)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Hospitalization | twelve months
  number of hospitalized days due to cardiac reasons
Six Minute Walk Test | day of discharge (approx. 5 - 10 days after operation)
  physical capacity expressed with the walking distance in meters

SECONDARY OUTCOMES:
Goal Attainment Scale (GAS) | three months
  level of attainment of individual goal: +2 = much more than expected, +1 = somewhat more than expected, 0 = goal achieved than expected, -1 = somewhat less than expected, -2 = much less than expected
Goal Attainment Scale (GAS) | twelve months
  level of attainment of individual goal: +2 = much more than expected, +1 = somewhat more than expected, 0 = goal achieved than expected, -1 = somewhat less than expected, -2 = much less than expected
HeartQoL | three months
  health-related quality of life; 14 items, min 0, max 42, higher scores indicating better health-related quality of life
HeartQoL | twelve months
  health-related quality of life; 14 items, min 0, max 42, higher scores indicating better health-related quality of life
Costs | up to 10 days
  direct costs in € associated with the operative procedure and the initial hospitalization using diagnosis related groups as classification system, in which diagnoses and treatments are valued according to their necessary economical expenditure

OTHER OUTCOMES:
European Health Literacy Questionnaire (HLS-EU-Q16) | day of discharge (approx. 5 - 10 days after operation)
  health literacy: 16 items, min 16, max 64, higher scores indicating lower health literacy
European Health Literacy Questionnaire (HLS-EU-Q16) | twelve months
  health literacy: 16 items, min 16, max 64, higher scores indicating lower health literacy
Brief Illnness Perception Questionnaire (BIPQ) | day of discharge (approx. 5 - 10 days after operation)
  individual concept of illness; 8 items, min 0, max 80, higher scores indicating worse illness perception
Brief Illnness Perception Questionnaire (BIPQ) | twelve months
  individual concept of illness; 8 items, min 0, max 80, higher scores indicating worse illness perception
Treatment Expectation Questionnaire (TEX-Q) | day of discharge (approx. 5 - 10 days after operation)
  treatment expectations; 15 items, min 0, max 150, higher scores indicating higher expectations of effects of the treatment
Treatment Expectation Questionnaire (TEX-Q) | three months
  treatment expectations; 15 items, min 0, max 150, higher scores indicating higher expectations of effects of the treatment
Treatment Expectation Questionnaire (TEX-Q) | twelve months
  treatment expectations; 15 items, min 0, max 150, higher scores indicating higher expectations of effects of the treatment
Patient Health Questionnaire-9 (PHQ-9) | day of discharge (approx. 5 - 10 days after operation)
  depressive symptoms; 9 items, min 0, max 27, higher scores indicating higher depressive symptoms
Patient Health Questionnaire-9 (PHQ-9) | three months
  depressive symptoms; 9 items, min 0, max 27, higher scores indicating higher depressive symptoms
Patient Health Questionnaire-9 (PHQ-9) | twelve months
  depressive symptoms; 9 items, min 0, max 27, higher scores indicating higher depressive symptoms
Generalized Anxiety Disorder-2 (GAD-2) | day of discharge (approx. 5 - 10 days after operation)
  anxiety symptoms; 2 items, min 0, max 6, higher scores indicating higher anxiety symptoms
Generalized Anxiety Disorder-2 (GAD-2) | three months
  anxiety symptoms; 2 items, min 0, max 6, higher scores indicating higher anxiety symptoms
Generalized Anxiety Disorder-2 (GAD-2) | twelve months
  anxiety symptoms; 2 items, min 0, max 6, higher scores indicating higher anxiety symptoms
Cardiac Anxiety Questionnaire (CAQ) | day of discharge (approx. 5 - 10 days after operation)
  cardiac anxiety; 17 items, min 0, max 68, higher scores indicating higher cardiac anxiety
Cardiac Anxiety Questionnaire (CAQ) | three months
  cardiac anxiety; 17 items, min 0, max 68, higher scores indicating higher cardiac anxiety
Cardiac Anxiety Questionnaire (CAQ) | twelve months
  cardiac anxiety; 17 items, min 0, max 68, higher scores indicating higher cardiac anxiety
Life Orientation Test - revised (LOT-R) | day of discharge (approx. 5 - 10 days after operation)
  optimism; 10 items, min 0, max 24, higher scores indicating higher optimism
Somatic Symptom Scale-8 (SSS-8) | day of discharge (approx. 5 - 10 days after operation)
  somatic symptom burden; 8 items, min 0, max 32, higher scores indicating higher somatic symptom burden
Somatic Symptom Scale-8 (SSS-8) | three months
  somatic symptom burden; 8 items, min 0, max 32, higher scores indicating higher somatic symptom burden
Somatic Symptom Scale-8 (SSS-8) | twelve months
  somatic symptom burden; 8 items, min 0, max 32, higher scores indicating higher somatic symptom burden
Somatic Symptom Disorder - B Criteria Scale (SSD-12) | day of discharge (approx. 5 - 10 days after operation)
  coping with somatic symptoms; 12 items, min 0, max 48, higher scores indicating worse coping with somatic symptoms
Somatic Symptom Disorder - B Criteria Scale (SSD-12) | three months
  coping with somatic symptoms; 12 items, min 0, max 48, higher scores indicating worse coping with somatic symptoms
Somatic Symptom Disorder - B Criteria Scale (SSD-12) | twelve months
  coping with somatic symptoms; 12 items, min 0, max 48, higher scores indicating worse coping with somatic symptoms
International Physical Activity Questionnaire Short Form (IPAQ) | day of discharge (approx. 5 - 10 days after operation)
  level of physical activity
International Physical Activity Questionnaire Short Form (IPAQ) | twelve months
  level of physical activity
Hand Dynamometer | day of discharge (approx. 5 - 10 days after operation)
  hand grip strength
Hand Dynamometer | twelve months
  hand grip strength
1 Minute Sit to Stand Test (1STS) | day of discharge (approx. 5 - 10 days after operation)
  physical capacity expressed with the number of repetitions
1 Minute Sit to Stand Test (1STS) | twelve months
  physical capacity expressed with the number of repetitions
Timed Up and Go (TUG) | day of discharge (approx. 5 - 10 days after operation)
  physical capacity expressed with the duration in seconds
Timed Up and Go (TUG) | twelve months
  physical capacity expressed with the duration in seconds
Six Minute Walk Test | twelve months
  physical capacity expressed with the walking distance in meters
Goal Attainment Scale (GAS) | day of discharge (approx. 5 - 10 days after operation)
  level of attainment of individual goal: +2 = much more than expected, +1 = somewhat more than expected, 0 = goal achieved than expected, -1 = somewhat less than expected, -2 = much less than expected
Readiness for Hospital Discharge Scale (RHDS) | day of discharge (approx. 5 - 10 days after operation)
  readiness for hospital discharge; 9 items, min 0, max 36, higher scores indicating higher readniss to discharge
5-level EQ-5D Health-related Quality of Life Questionnaire (EQ-5D-5L) | three months
  health-related quality of life; 6 items, interpretation following an algorythm between 1 (best possible health condition) and <0 (worst possible health condition)
5-level EQ-5D Health-related Quality of Life Questionnaire (EQ-5D-5L) | twelve months
  health-related quality of life; 6 items, interpretation following an algorythm between 1 (best possible health condition) and <0 (worst possible health condition)
Questionnaire for Health-Related Resource Use in an Elderly Population (FIMA) | twelve months
  use of health care services; 11 items collecting numbers of health care services and days of usage, min 0, higher scores indicating higher usage of services

CONTACTS AND LOCATIONS:
Overall Officials: Evaldas Girdauskas, Prof., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - Universitätsklinikum Augsburg, Augsburg, Bavaria
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kubitz JC, Schulte-Uentrop L, Zoellner C, Lemke M, Messner-Schmitt A, Kalbacher D, Sill B, Reichenspurner H, Koell B, Girdauskas E. Establishment of an enhanced recovery after surgery protocol in minimally invasive heart valve surgery. PLoS One. 2020 Apr 9;15(4):e0231378. doi: 10.1371/journal.pone.0231378. eCollection 2020. PMID 32271849
- [Background] Petersen J, Kloth B, Konertz J, Kubitz J, Schulte-Uentrop L, Ketels G, Reichenspurner H, Girdauskas E. Economic impact of enhanced recovery after surgery protocol in minimally invasive cardiac surgery. BMC Health Serv Res. 2021 Mar 20;21(1):254. doi: 10.1186/s12913-021-06218-5. PMID 33743698
- [Background] Klotz SGR, Ketels G, Behrendt CA, Konig HH, Kohlmann S, Lowe B, Petersen J, Stock S, Vettorazzi E, Zapf A, Zastrow I, Zollner C, Reichenspurner H, Girdauskas E. Interdisciplinary and cross-sectoral perioperative care model in cardiac surgery: implementation in the setting of minimally invasive heart valve surgery (INCREASE)-study protocol for a randomized controlled trial. Trials. 2022 Jun 23;23(1):528. doi: 10.1186/s13063-022-06455-x. PMID 35739541
- See also: summary of the project on the sponsor's website — https://innovationsfonds.g-ba.de/projekte/neue-versorgungsformen/increase-interdisziplinaere-und-sektorenuebergreifende-versorgung-in-der-herzchirurgie-am-beispiel-von-minimal-invasiven-herzklappeneingriffen.377